CLINICAL TRIAL: NCT06267794
Title: Double-blind Clinical Trial to Evaluate the Safety and Efficacy of Two Doses of Prolonged Release Pirfenidone, Compared Against Placebo Plus Conventional Therapy in Patients With Compensated Liver Cirrhosis.
Brief Title: Prolonged Release Pirfenidone Versus Placebo in Compensated Cirrhosis.
Acronym: ODISEA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jorge L Poo (Other)
Responsible Party: Sponsor-Investigator, Jorge L Poo, PROMHEPA administrator and Co-Investigator, Grupo Mexicano para el Estudios de las Enfermedades Hepaticas
Organization: Grupo Mexicano para el Estudios de las Enfermedades Hepaticas (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ODISEA Study
Record Dates: First submitted 2024-01-22; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Liver Fibrosis; Cirrhosis, Liver; Chronic Liver Disease
Keywords: Liver fibrosis; Fibrosis treatment; Fibrosis reversibility; Pirfenidone; Prolonged release pirfenidone
MeSH Terms: conditions — Liver Cirrhosis | interventions — pirfenidone

STUDY DESIGN:
Intervention Model Description: Double blind, placebo-controlled multicenter study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Placebo will be identical to medication.
  Methods to assign treatment:
  Before assigning numbers to subjects, the researcher must confirm that the inclusion criteria have been met, that none of the exclusion criteria apply, that written and signed informed consent has been obtained, that the evaluations of the scrutiny (of admission) and that the required laboratory results are available and meet the admission criteria. To do this, the centers will be assisted with a check list format that contains all the selection criteria.
  The person responsible for the medication at the research site will contact the Randomization center, where the treatment will be assigned to the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Prolonged release pirfenidone (PR-PFD), 1200 mg group (Experimental): Subjects will receive one tablet during breakfast and 2 tablets during dinner.
  Interventions: Drug: Pirfenidone 1200 mg
- PR-PFD, 1800 mg group (Active Comparator): Subjects will receive one tablet during breakfast and 2 tablets during dinner.
  Interventions: Drug: Pirfenidone 1800 mg
- Placebo group (Placebo Comparator): Subjects will receive one tablet during breakfast and 2 tablets during dinner.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pirfenidone 1200 mg — 1200 mg dosage. Additionally, all participating subjects will receive standard treatment care for patients with cirrhosis.
  Other Names: Prolonged-release pirfenidone
  Arms: Prolonged release pirfenidone (PR-PFD), 1200 mg group
Drug: Pirfenidone 1800 mg — 1800 mg dosage. Additionally, all participating subjects will receive standard treatment care for patients with cirrhosis.
  Other Names: Prolonged-release pirfenidone
  Arms: PR-PFD, 1800 mg group
Drug: Placebo — 0 mg dosage. Additionally, all participating subjects will receive standard treatment care for patients with cirrhosis.
  Arms: Placebo group

SUMMARY:
This will be a multicenter, double-blind clinical trial to evaluate the safety and efficacy of two doses of prolonged release pirfenidone, compared against placebo plus conventional therapy in patients with compensated liver cirrhosis. The study will be conducted in compliance with International Standard good clinical practices (GCPs) and the Declaration of Helsinki. The protocol is approved by a local Institutional Review Board and registered in clinical trials.gov.

DETAILED DESCRIPTION:
Liver cirrhosis represents a clear public health problem all over the world. In Mexico it ranks sixth as a cause of general mortality (third place in men and seventh in women) with 28,000 to 30,000 deaths per year, according to the latest National Institute of Statistics and Geography report. and the National Population Council.

Hepatic stellate cells are, to date, the main fibrogenic cells in the liver, thus becoming one of the most important therapeutic targets for treatment. Advances in the understanding of the molecular biology of the liver have allowed us to devise therapeutic strategies in order to avoid fibrosis and the consequent loss of liver function.

In 1994, a preliminary report was released publishing the antifibrotic properties of Pirfenidone (5-methyl-1-phenyl-2-[1H]-pyridone, here and after PFD), a drug initially known for its analgesic and anti-inflammatory capabilities.

In 1995, its antifibrotic properties were described when administered in a hamster model with pulmonary fibrosis induced by bleomycin. Its mechanism of action was not completely well established at that time. It was known to be at the transcriptional level and was shown to modulate the deposition of extracellular matrix, the production of cytokines, growth factors and fibroblast proliferation. It is associated with the inhibition of the production and activity of tumor necrosis factor (TNF-α), transforming growth factor (TGF-ß), interferon-gamma and interleukin (IL) -6 and increases the production of anti-inflammatory cytokines such as IL-10.

The PFD molecule has shown promising effects both in vitro and in vivo in the prevention and treatment of idiopathic pulmonary fibrosis (IPF), in the prevention of capsular contracture after breast implants, renal interstitial fibrosis, in particular focal and segmental glomerulosclerosis or diabetic nephropathy and a wide range of conditions that share the phenomenon of abnormal scarring including hypertrophic and keloid scars, peritoneal adherences, neurofibromatosis and uterine fibromyomas. More recently it has also been evaluated in secondary and progressive variety multiple sclerosis, with promising results. In IPF, PFD has been positioned as the standard of care because it improves the outcomes, slowing down or blocking the decline of respiratory function and improving survival.

In models of liver fibrosis, PFD has also been shown to have antifibrotic activity. In experimental cirrhosis models in rats, it has been found that PFD decreases the levels of aminotransferases and bilirubins and stimulates cell regeneration. At the molecular level, a considerable decrease was also observed in the expression of pro-fibrogenic genes such as collagen I, III and IV, TGF ß-1, Smad-7, tissue inhibitor of metalloproteinases (TIMP-1) and plasminogen inhibitor 1 (PAI-1). In this way, it is known that PFD has various anti-inflammatory and antifibrotic properties, which have molecular support for its application as a potential treatment for liver cirrhosis.

Since 2000, the Mexican company Grupo Medifarma has manufactured the molecule 1-phenyl-5-methyl-2- (1H)-pyridone (PFD), hereinafter KitosCell ® LP in its plant located in Jiutepec, Morelos. Formulation details are confidential and protected by patent rights. However, the pharmacological components of the product are balanced and in sufficient concentration to achieve a stable product with homogeneous concentrations in the production batches. The stability of the KitosCell ® LP formula has been tested from a biochemical, biological and physical point of view. Additionally, the in vitro dissolution tests resulted within the expected physiological concentrations, as well as the sterility tests required by the Mexican Pharmacopeia. From a production point of view, Grupo Medifarma has the experience to demonstrate adherence to good manufacturing practices of the product under study in accordance with the requirements of the Ministry of Health.

Molecular biology studies have established that the mechanism of action of PFD is carried out at the transcriptional level, in the place where an interface occurs between the signals of specific genes or group of genes, which are being transmitted to the process by the following factors:

NF = transcriptional factor regulating the expression of proinflammatory genes. AP1 = a transcriptional factor that regulates expression of collagen proteins.

For all these reasons, PFD is considered a therapeutic resource for:

* Prevent the formation of fibrotic lesions.
* Reduce pre-existing fibrotic progression.
* Reverse fibrotic lesions.

As preclinical studies, studies were carried out in experimental models of cirrhosis in rats. There were 3 groups of rats: 1 control group and 2 groups with different doses of PFD (200 mg and 500 mg) per day, for 11 weeks. They were subsequently sacrificed and histopathological analysis of the liver showed a significant decrease in liver fibrosis in the groups that received PFD.

The first pilot clinical study to evaluate the effect of pirfenidone in patients with viral C liver fibrosis was carried out by J. Armendáriz-Borunda et al., at the Civil Hospital of Guadalajara in conjunction with the Institute of Molecular Biology in Medicine and Gene Therapy.

In this open pilot study, only 15 patients with liver fibrosis of various etiologies and different liver functional stages were included. Liver biopsies performed after 12 months suggested that in 53.3% of patients there was a reduction of two points or more in the necro-inflammatory index (HAI), 60% of steatosis decreased and 30% of fibrosis improved, while 70% regeneration activity was detected.

Problem Statement.

The present study aims to evaluate the efficacy, safety and pharmacodynamics of a formulation based on prolonged release Pirfenidone ( KitosCell® LP) , prepared by Grupo Medifarma, in two dosages (1200 mg and 1800 mg) vs. placebo plus conventional treatment for patients. with liver cirrhosis in the compensated phase with Child-Pugh functional class A and B (≤8 points) without a history of previous complications, of different causes .

The clinical tests aim to cover the international requirements for the development of a new drug under study (phases 1, 2 and 3) with antifibrotic effect. Therefore, if the safety and then the effectiveness of the product are demonstrated, a new therapeutic strategy can be offered for this complex health problem.

Justification of the Study.

Liver cirrhosis is the fifth cause of general mortality in our country, with around 28,000 deaths each year. To date, there is no proven effective therapy that allows reversing or inhibiting the fibrogenic process. This complex disease impacts the economically active population, causing great losses by causing work incapacity as well as the morbidity and mortality that it entails. The investigators consider that it is desirable to carry out a study, with a controlled and double-blind design that allows us to provide new knowledge of the efficacy and safety of the drug under study, in accordance with the recently published recommendations of the American Association for the Study of Liver Diseases (AASLD). by Natalie J. Torok and collaborators (Jan 27, 2015).

ELIGIBILITY:
Inclusion Criteria:

1. Both genders over 18 years of age.
2. Patients with clinical, biochemical, radiological diagnostic confirmation as well as evidence of grade 4 fibrosis based on an invasive (liver biopsy) or non-invasive method (fibrotest and/or fibroscan).
3. With functional class A (score of 5 and 6) and B (score of 7 or 8) on the Child-Pugh scale.
4. Optionally, transjugular liver biopsy with measurement of the portal system flow pressure gradient, in at least 20% of the population.
5. Be controlled with medications that are consumed at stable doses for at least 30 days.
6. Have a BMI greater than 19.1 kg/m 2 and less than 34.9 kg/m 2
7. Have the required standardized and homogeneous diet for patients
8. Do not drink alcoholic beverages for at least one year prior to the start of the study.
9. Electrocardiogram normal or without clinical significance.
10. Laboratory tests that confirm your condition and functional class, with results that, in the opinion of the principal investigator, do not put the patient at risk:

    1. Complete blood count, with hemoglobin values ≥ 12 g/dL, leukocytes ≥ 3,500 mL, platelets ≥ 50,000 mL
    2. Blood chemistry (glucose, urea, creatinine, uric acid, cystatin C).
    3. Complete liver function tests (total protein, globulin, albumin, ALT, AST, gamma-glutamyltransferase (GGT), alkaline phosphatase (AP), lactic dehydrogenase (LDH), Total Bilirubin, C-reactive Protein).
    4. Fibrotest and/or FibroScan with a result of F4.
    5. General urine examination.
11. Inclusion Criteria for patients with hepatitis C virus liver damage.

    1. Having been previously treated with standardized antiviral management
    2. More than 12 months have passed since the end of antiviral treatment.
12. Inclusion Criteria for patients with liver damage of autoimmune etiology.

    a. Be under immunosuppressive treatment (steroid plus azathioprine) at a stable dose for at least 6 months at the beginning of the study.
13. Inclusion Criteria for patients with liver damage due to alcohol.

    1. With alcohol inactivity for at least one year before the start of the study.

Exclusion Criteria:

1. Pregnancy and breastfeeding.
2. History of known allergy or hypersensitivity to PFD.
3. Have liver cirrhosis with functional reserve B (score of 9) or functional reserve C (score of 10 or more) on the Child-Pugh scale. 11 (See annexes).
4. History of Upper Gastrointestinal Bleeding, Ascites, Hepatic Encephalopathy or any other complication due to previous Portal Hypertension.
5. Body Mass Index less than 19 kg/m 2 or greater than 35 kg/m 2
6. Hemoglobin values less than 12 g/dL.
7. Have participated in another clinical study in the 60 days prior to the start of this one.
8. Hospitalization within 30 days prior to the start of medication administration.
9. Concomitant systemic infection other than hepatitis C virus (HCV), including Respiratory Tract Infections , Urinary Tract Infections, human immunodeficiency virus (HIV), cellulitis, etc.
10. Current use (less than 1 month) of colchicine, ursodeoxycholic acid, silimarin, or s-adenosine methionine, or cytotoxic agent, cytokine modulator or receptor antagonist, daily sildenafil or fluvoxamine, theophylline or other methylxanthines, or alternative medicine.
11. Have clinical data of pulmonary fibrosis, heart, respiratory or kidney failure (serum creatinine > 1.5 mg/dL).
12. Other medications that, in the opinion of the principal investigator, may interfere with the study.
13. Any other clinical condition that causes fibrosis other than liver fibrosis or a condition that, in the opinion of the principal investigator, could compromise the safety and well-being of the patient or put the conduct of the study at risk, such as hepatocellular carcinoma.

Elimination criteria

Any patient who presents a clinical finding compatible with decompensated cirrhosis (bleeding of variceal origin, clinical ascites, evident hepatic encephalopathy, hepatocellular carcinoma) or an adverse event or condition that, in the opinion of the principal investigator, warrants suspension of the patient's participation will be suspended from the study, but their data will be considered in the "intention to treat" analysis, when applicable.

In the event that a serious adverse event occurs that, in the opinion of the principal investigator, warrants suspension of the patient's participation. In these cases, clinical and biochemical data will be considered in the intention-to-treat analysis, when applicable.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-06-26 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Change in liver fibrosis | 6, 12, 18 and 24 months
  Fibrosis change based on Hepatic Elastography.
  Variation of fibrosis score by at least 30% in kilo Pascals (kPa) according to accurate hepatic elastography measurements.
  Fibrosis change based on Fibrotest. Change of fibrosis score by at least 10% in Fibrotest units.
Clinical side effects | 6, 12, 18 and 24 months
  Clinical side effects will be evaluated according to World Health Organization guidelines.
  The following definitions will be used to grade the severity of adverse events:
  Mild: Awareness of sign, symptom or event, but easily tolerated. Moderate: Discomfort sufficient to cause interference with usual activity and may require intervention.
  Serious: Disabling without ability to do usual activities, or significantly affects clinical status and requires intervention.
  Puts Life at Risk: Immediate risk of death (Sponsor must be notified within 24 hours).
  The Investigators must also evaluate the relationship of any adverse event with the use of the study drug, based on the available information, according to the following guidelines:
  0 = Unrelated
  1. = Possibly related
  2. = Probably related

SECONDARY OUTCOMES:
Improvement in Child Pugh score | 6, 12, 18 and 24 months
  Change in Child Pugh score. Variations of at least one point compared to baseline values.
  In Hepatology, the Child-Pugh score is used to evaluate the prognosis of chronic liver disease, mainly cirrhosis. Although it was originally used to predict mortality during liver surgery, it is also useful for a patient's prognosis.
  The score employs five clinical measures of liver disease: bilirubin, albumin, prothrombin time, ascites and encephalopathy. Each measure is scored 1-3, with 3 indicating most severe derangement.
  Chronic liver disease is classified into Child-Pugh class A to C, employing the following criteria:
  Child Pugh A: 5-6 points Child-Pugh B; 7-9 points Child Pugh C: 10-15 points
Improvement in MELD score | 6, 12, 18 and 24 months
  Change in participants's model for end-stage liver disease (MELD) score Variations of at least one point compared to baseline values.
  MELD score estimates a patient's chances of surviving their disease over the next three months of life and ranges from six to 40 and is based on results from several lab tests. The higher the number, the more likely participants are to receive a liver from a deceased donor when an organ becomes available.
  MELD score is based on results from four blood tests that, together, show how well participants' body is functioning.
  Prothrombin time as international normalized ratio (INR): Indicates whether participant´s liver is making the proteins necessary for blood to clot.
  Creatinine: Indicates how well participant´s kidneys are working. Bilirubin: Indicates how well participant´s liver is clearing a substance called bile.
  Serum sodium: Indicates how well participants' body is regulating fluid balance.
Improvement in bilirrubin and albumin | 6, 12, 18 and 24 months
  Improvement in Liver function values: bilirubin Improvement by at least 30% in serum Bilirubin levels (mg/dL)
  Improvement in Liver function values: albumin Improvement by at least 30% in serum albumin levels (mg/dL)
Improvement in prothrombin time | 6, 12, 18 and 24 months
  Improvement in Liver function values: prothrombin time Improvement by at least 30% in INR values.
Improvement in liver enzymes | 6, 12, 18 and 24 months
  Improvement in transferases values: alanine aminotransferase (ALT) Improvement by at least 30% in enzyme values (IU/L)
  Improvement in transferases values: aspartate aminotransferase (AST) Improvement by at least 30% in enzyme values (IU/L)
Improvement in EuroQol Visual analog scales | 6, 12, 18 and 24 months
  1. Improvement in the quality of life self-assessment scale with the Visual EuroQol scale.
  The scale ranges from 0 (worst imaginable health state) to 100 (best imaginable health state).
Improvement in EuroQol five dimensions Scale | 6, 12, 18 and 24 months
  The descriptive system includes five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Their responses are coded as a number (1, 2, or 3) corresponding to the respective level of severity: 1 indicates no problems, 2 some problems, and 3 extreme problems. In this way, a person's health status profile can be defined by a 5-digit number, ranging from 11111 (having no problems in any of the dimensions) to 33333 (having extreme problems in all dimensions). Finally, each patient receives a score with an index ranging from 1 to 0. The maximum quality of life values would be 1. The index could also be scored between 0 and 100%.
Improvement in modified fatigue impact scale (MFIS) | 6, 12, 18 and 24 months
  Fatigue is a feeling of physical tiredness and lack of energy that many people experience from time to time.
  Items on the MFIS can be aggregated into three subscales (physical, cognitive, and psychosocial), as well as into a total MFIS score.
  The total MFIS score can range from 0 to 84. It is computed by adding scores on the physical, cognitive, and psychosocial subscales. All items are scaled so that higher scores indicate a greater impact of fatigue on a person's activities.